CLINICAL TRIAL: NCT07073729
Title: Corneal Neurotization: A Study on the Outcomes of Nerve Repair for Corneal Sensory Dysfunction
Brief Title: Corneal Neurotization vs. Cenergermin for Neurotrophic Keratitis: A Pilot Study
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: London Health Sciences Centre Research Institute OR Lawson Research Institute of St. Joseph's (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CamachoNK2025
Record Dates: First submitted 2025-07-09; First posted 2025-07-18 (Actual); Last update posted 2025-07-18 (Actual); Status verified 2025-06

CONDITIONS: Neurotrophic Keratitis
Keywords: Corneal Neurotization; Cenergermin; Neurotrophic Keratopathy; Corneal Sensory Dysfunction
MeSH Terms: interventions — cenegermin

STUDY DESIGN:
Intervention Model Description: Participants will receive either corneal neurotization surgery or Cenergermin (Oxervate) eye drops based on their clinical care plan. No randomization is used. The study will follow both groups over a 12-month period.
Masking Description: No masking is used in this feasibility study. All parties are aware of the intervention received.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Corneal Neurotization (Experimental): Participants in this arm will receive corneal neurotization surgery as part of their standard clinical care. The surgical procedure involves transferring healthy donor nerves to the anesthetic cornea in order to restore corneal sensation. Participants are followed over 12 months without randomization.
  Interventions: Procedure: Corneal Neurotization
- Cenergermin (Active Comparator): Participants in this arm will receive topical Cenergermin (Oxervate) eye drops, a recombinant human nerve growth factor approved for treatment of neurotrophic keratitis. Treatment is selected based on clinical decision-making. Participants are followed over 12 months as part of routine care.
  Interventions: Drug: Cenergermin

INTERVENTIONS:
Procedure: Corneal Neurotization — Surgical technique involving the transfer of healthy donor sensory nerves to the anesthetic cornea to restore corneal innervation and sensation in patients with neurotrophic keratitis.
  Other Names: Corneal Nerve Transfer; Corneal Sensory Nerve Grafting
  Arms: Corneal Neurotization
Drug: Cenergermin — Topical recombinant human nerve growth factor (rhNGF) approved for the treatment of neurotrophic keratitis. Administered as eye drops, it promotes epithelial healing and nerve regeneration.
  Other Names: Oxervate
  Arms: Cenergermin

SUMMARY:
This pilot study evaluates the feasibility and outcomes of two treatment approaches for corneal sensory dysfunction due to neurotrophic keratitis (NK): corneal neurotization surgery and topical Cenergermin (Oxervate). Participants will receive treatment based on clinical decision-making, not randomization, and will be followed for 12 months through eight visits at the Ivey Eye Institute, St. Joseph's Health Care London. Data collected during routine eye examinations and validated quality-of-life questionnaires will be used to assess visual outcomes, corneal structure and function, and patient-reported well-being. This feasibility study is funded by the Lawson Research Institute Internal Research Fund and is intended to generate preliminary evidence for a future randomized trial.

DETAILED DESCRIPTION:
Neurotrophic keratitis (NK) is a rare, progressive condition characterized by impaired corneal sensation and reduced nerve function. It affects approximately 5 in 10,000 individuals worldwide and more than 6,000 Canadians annually. If untreated, NK can lead to corneal scarring, ulceration, and irreversible vision loss. Two existing treatments are currently in use: corneal neurotization, a surgical technique that transfers healthy donor nerves to the cornea and topical Cenergermin (Oxervate), a recombinant human nerve growth factor that promotes epithelial healing and nerve regeneration.

This single-center, prospective pilot study is designed to assess the feasibility of conducting a larger comparative trial between these two treatment approaches. Specifically, the study will determine whether it is clinically and logistically feasible to compare outcomes between patients undergoing neurotization surgery and those receiving Cenergermin drops as part of their standard care.

Ten adult participants (aged ≥19) with moderate to severe NK will be recruited from the Ivey Eye Institute at St. Joseph's Health Care London. Participants will receive either surgical or medical treatment based on standard clinical care decisions. No additional interventions will be introduced for research purposes.

Participants will be followed across eight time points: baseline (before treatment), 1 day, 1 week, 1 month, 3 months, 6 months, 9 months, and 12 months. Each visit will include routine clinical evaluations such as corneal sensitivity testing, corneal nerve imaging, slit lamp exams, intraocular pressure, visual acuity and contrast testing, and a brief quality-of-life questionnaire.

All data will be collected through standard, non-invasive assessments during regular clinical follow-up. There will be no masking; both participants and clinicians will be aware of the assigned treatment.

This research is part of a pilot grant funded by the Lawson Health Research Institute and will provide critical data to inform the development of a larger, fully powered randomized controlled trial.

ELIGIBILITY:
Inclusion Criteria:

* Adults aged 19 years and older.
* Diagnosis of neurotrophic keratitis with reduced or absent corneal sensation.
* Clinical indication for either corneal neurotization surgery or topical Cenergermin treatment, as determined by the treating ophthalmologist.
* Ability to provide informed consent.

Exclusion Criteria:

* Active ocular infection or inflammation.
* Previous corneal neurotization procedure in the affected eye.
* Contraindications to general anesthesia or surgical intervention.
* Participation in another interventional clinical trial within the past 3 months.

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Estimated)
Dates: Start 2025-08-01 (Estimated); Primary Completion 2026-08-01 (Estimated); Study Completion 2027-08-01 (Estimated)

PRIMARY OUTCOMES:
Change in Corneal Sensitivity | Baseline and 12 months post-treatment
  Measured using Cochet-Bonnet esthesiometry to evaluate restoration of corneal sensation following intervention.

SECONDARY OUTCOMES:
Change in best-corrected visual acuity | Baseline and 12 months post-intervention
  Best-corrected visual acuity will be assessed using a standardized Snellen chart or equivalent method. The goal is to evaluate visual improvement following corneal neurotization or cenergermin treatment.
Overall Impact of the Procedure | 12 months
  Comprehensive assessment of the overall effects of corneal neurotization, including clinical and functional outcomes as well as patient-reported measures of ocular comfort, perceived visual function, and general well-being at 12 months post-procedure.

CONTACTS AND LOCATIONS:
Overall Officials: Alex Camacho, MD, MSc, Principal Investigator — Western University, Ophthalmology; Cindy Hutnik, MD, PhD, Department Chief, Study Chair — Western University, Ophthalmology; Monali Malvankar, PhD, Professor, Study Chair — Western University, Ophthalmology; Anastasiya Vinokurtseva, MD, Resident, Study Chair — Western University, Ophthalmology
Locations (1):
- Ivey Eye Institute, St. Joseph's Health Care London, London, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No
The plan to share individual participant data (IPD) is currently under consideration and will depend on future institutional policies, data privacy constraints, and the outcomes of the study.